CLINICAL TRIAL: NCT03034616
Title: in Vivo Activation of Ovarian Cortex in Premature Ovarian Insufficiency
Brief Title: Ovarian Laparoscopic In Vivo Activation of Ovary for Premature Ovarian Insufficiency
Acronym: OLIVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ariel Revel, Principal investigator, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 029416
Record Dates: First submitted 2017-01-13; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Primary Ovarian Insufficiency
Keywords: Primary ovarian insufficiency; In-vivo activation
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ex vivo activation (Experimental): 'OLIVA device' in patients that undergo oophorectomy on the cortex of the removed ovary we will perform 5 parallel slashes 3 cm long.
  this will be followed by investigation by the pathologist as to the depth of cuts.
  Interventions: Device: OLIVA device
- in vivo activation (Active Comparator): 'OLIVA device' in patients undergoing oophorectomy before the resection from is pedicle on cortex of the ovary we will perform 5 parallel slashes 3 cm long. following oophorectomy investigation by the pathologist as to the depth of cuts and proximity to blood vessels.
  Interventions: Device: OLIVA device
- POI OLIVA (Active Comparator): 'OLIVA device' in patients with premature ovarian failure and following safety data from arm 2 activation by ovarian slashing will be performed laparoscopically by closed cutting device (OLIVA). follow-up by sonography and hormonal markers of ovarian activity
  Interventions: Device: OLIVA device

INTERVENTIONS:
Device: OLIVA device — OLIVA device is a laparoscopic device with a standard handle and a tip built of 5 parallel razor blades enclosed by protective cap opened by a separate button.
  This device will enable to perform shallow slashes on the ovarian cortex following the grasping of the ovary without damaging other abdominal and pelvic organs

SUMMARY:
The OLIVA device will enable to perform shallow slashes on the ovarian cortex in patients undergoing oophorectomy. Prior to the resection of the ovary from the pedicle we will perform 5 parallel slashes 3 cm long. following oophorectomy investigation by the pathologist as to the depth of cuts and proximity to blood vessels and later.

DETAILED DESCRIPTION:
The OLIVA device is built of 5 parallel razor blades enclosed by protective cap

ELIGIBILITY:
Inclusion Criteria:

* Peri/menopausal women undergoing laparoscopic oophorectomy

Exclusion Criteria:

* Women with ovarian malignancy
* Women with polycystic ovarian syndrome

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Depth of cuts and closeness to blood vessel | Up to 30 days after procedure
  The pathologist will measure the ovarian tissue after oophorectomy. The pathologist will assess whether the cuts into the cortex are superficial or penetrating the cortex into the medulla of the ovary. Another assessment is proximity of the cuts to ovarian vessels. The pathology report will aggregate the results of all measurements and will assess the safety of the OLIVA device

SECONDARY OUTCOMES:
Proximity of cuts to blood vessel | Up to 30 days after procedure
  The pathologist will measure the ovarian tissue after oophorectomy. The pathologist will assess whether the cuts into the cortex are superficial or penetrating the cortex into the medulla of the ovary. Another assessment is proximity of the cuts to ovarian vessels. The pathology report will aggregate the results of all measurements and will assess the safety of the OLIVA device

IPD SHARING:
Plan to Share IPD: No